CLINICAL TRIAL: NCT01294891
Title: Microvascular and Cardiac Dysfunction in Paroxysmal Nocturnal Hemoglobinuria and Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Other Study IDs: IRB00006948
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Rheologic Disease; Sickle Cell Disease; Paroxysmal Nocturnal Hemoglobinuria
Keywords: Rheology; Sickle cell; Paroxysmal nocturnal hemoglobinuria; contrast ultrasound
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinuria, Paroxysmal | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: Age matched healthy subjects
  Interventions: Other: Imaging
- Sickle Cell Patients: Patients with established SCD
  Interventions: Other: Imaging
- Paroxysmal Nocturnal Hemoglobinuria patients: Patients with PNH
  Interventions: Other: Imaging

INTERVENTIONS:
Other: Imaging — Contrast ultrasound perfusion imaging and complete echocardiography

SUMMARY:
The purpose of this study is to examine how abnormal blood flow in the small vessels (microvessels) of the heart, muscle and kidney in paroxysmal nocturnal hemoglobinuria (PNH) or sickle cell disease leads to poor functioning of the heart and kidney. To test this question, the investigators will perform imaging tests (contrast ultrasound perfusion imaging) to look at the flow and function of these microvessels and compare this information to heart and kidney function. To further look at this question, patients who have PNH will be studied before and after starting a new drug (Soliris) that decreases damage to blood cells. In patients with sickle cell disease, patients will be studied at baseline (not during a pain crisis) and also during a pain crisis if one develops.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of PNH or SCD Age > 18 years old

Exclusion Criteria:

* Pregnant or lactating women Presence of significant right to left shunting Allergy to ultrasound contrast agent Reactive airways disease Significant peripheral or coronary artery disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with SCD or PNH who are seen in the OHSU Hematology clinic and are asked to participate
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Microvascular perfusion | 1 hour
  1. Myocardial microvascular blood flow (MBF) and capillary blood velocity (CBV) on study day.
  2. Renal MBF on study day
  3. Skeletal muscle MBF and CBV on study day
  4. Myocardial MBF and CBV during hyperemia
  5. Skeletal muscle CBV during hyperemia

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States